CLINICAL TRIAL: NCT03338686
Title: A Prospective Randomized Clinical Trial to Compare Free Gingival Grafts and Connective Tissue Grafts Around Implants With Lack of Keratinized Mucosa
Brief Title: To Compare Free Gingival Grafts and Connective Tissue Grafts Around Implants With Lack of Keratinized Mucosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Ramzi V. Abou-Arraj, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STS-15
Record Dates: First submitted 2017-10-03; First posted 2017-11-09 (Actual); Results first posted 2021-04-08 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-08

CONDITIONS: Dental Implants; Alveolar Mucosa
Keywords: Keratinized tissue; Keratinized mucosa; Attached mucosa; Dental implants; Free gingival graft; Connective tissue graft; Patient-centered outcomes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Free Gingival Graft (Active Comparator): Free Gingival Graft (FGG)
  Interventions: Procedure: Free Gingival Graft (FGG)
- Connective Tissue Graft followed by Laser Gingivoplasty (Experimental): Connective Tissue Graft (CTG) followed by Laser Gingivoplasty
  Interventions: Procedure: Connective Tissue Graft followed by Laser Gingivoplasty

INTERVENTIONS:
Procedure: Free Gingival Graft (FGG) — Free Gingival Graft (FGG) was performed on all study sites in this arm.
  Other Names: palatal autogenous soft tissue graft
  Arms: Free Gingival Graft
Procedure: Connective Tissue Graft followed by Laser Gingivoplasty — Connective Tissue Graft followed by Laser Gingivoplasty one month later on all study sites in this arm.
  Other Names: palatal autogenous subepithelial soft tissue graft
  Arms: Connective Tissue Graft followed by Laser Gingivoplasty

SUMMARY:
This study will compare two commonly used soft tissue grafting techniques (free gingival graft, FGG vs. connective tissue graft, CTG) to augment the soft tissue around dental implants with a lack of keratinized mucosa.

To investigators knowledge, these 2 types of grafts have not been compared for differences in clinical (amount of KM increase, tissue thickness increase and esthetics) and patient-centered outcomes (pain, swelling, change in daily activities) in a controlled study.

DETAILED DESCRIPTION:
Research data and daily clinical observations reveal that implants with lack of surrounding keratinized mucosa KM (gingiva-like tissue that normally surrounds natural teeth) are more prone to persistent gingival inflammation, faster disease progression and compromised plaque control. Soft tissue grating (with FGG or CTG) aims at changing the nature of peri-implant soft tissue by creating or increasing the zone of keratinized mucosa (KM) surrounding implants in question. While FGG is typically associated with higher postoperative discomfort than CTG, it has also been considered the gold standard in the treatment of these clinical conditions.

Specific aims for this project include the evaluation of:

* KM width at 6 and 12 months following grafting with FGG and CTG
* Change in tissue thickness of the grafted sites at 6 and 12 months
* Esthetic outcomes using a newly developed peri-implant esthetic scale at 6 and 12 month
* Patient centered outcomes including pain, bleeding, swelling and change in daily activities at 1 week for both groups and at 1 month for the CTG group

ELIGIBILITY:
Inclusion Criteria:

1. English speaking
2. At least 18 years old
3. Must be a patient of the UAB Dental School, able to read and understand informed consent document
4. One or more adjacent dental implants having <2mm in width of keratinized mucosa or attached mucosa <1mm around their buccal aspect Contra-lateral or opposing implant sites with above criteria may be included and randomly assigned to soft tissue graft type
5. No crestal bone loss or minimal bone resorption not extending apical to first implant thread
6. Presence of periodontally healthy neighboring teeth, healthy implants or edentulous ridge on either side of the involved site (s)
7. Implants requiring soft tissue grafting after placement (>2 months): implants with healing abutments awaiting restoration or after delivery of temporary/permanent restoration

Exclusion Criteria:

1. Non-English speaking
2. Less than 18 years old
3. Smokers/tobacco users (>10 cigarettes/day)
4. Patients with systemic pathologies or conditions contraindicating oral surgical procedures or adversely affecting wound healing
5. Presence of peri-implantitis, acute infection and/or suppuration at the implant placement site (s)
6. Presence of soft tissue recession exposing threads at implant site
7. Presence of bony dehiscence at implant site (s)_ at time of surgery
8. Previous soft tissue grafting at the implant site (s)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-01-07 (Actual); Primary Completion 2018-10-09 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramzi V Abou-Arraj, DDS, MS, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, School of Dentistry, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomization was performed by site in the mouth (dental implant) to receive either FGG intervention or CTG intervention. As a result, some participants received only one of the 2 interventions if they only had one qualifying site (=dental implant) while other participants received both interventions if they had multiple implants that met the inclusion criteria. Total FGG implant sites=14, total CTG sites=12.
Units Other Than Participants: implants
Groups:
- FGG + CTG: Both FGG and CTG (at different implants in the same patient)
Period: Overall Study
Arm/Group | Free Gingival Graft | Connective Tissue Graft Followed by Laser Gingivoplasty | FGG + CTG
Started | 2; 2 implants | 5; 5 implants | 7; 19 implants (12 FGG implant sites and 7 CTG implant sites for this Arm/Group)
Completed | 2; 2 implants | 5; 5 implants | 7; 19 implants
Not Completed | 0; 0 implants | 0; 0 implants | 0; 0 implants

BASELINE CHARACTERISTICS:
Units Other Than Participants: implants
Groups:
- Total: Total of all reporting groups
Arm/Group | Free Gingival Graft | Connective Tissue Graft Followed by Laser Gingivoplasty | FGG + CTG | Total
Number analyzed (Participants) | 2 | 5 | 7 | 14
Number analyzed (implants) | 2 | 5 | 19 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 3 | 5 | 8
  >=65 years | 2 | 2 | 2 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 5 | 11
  Male | 1 | 0 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 0 | 4
  White | 1 | 2 | 7 | 10
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Increase in Keratinized Mucosa (in mm) Between the Two Grafts
Description: Compare the increase in keratinized mucosa (KM) between two commonly used soft tissue grafting techniques (FGG and CTG) by quantifying KM widths (in mm) at 12 months following soft tissue grafting.
Time Frame: From baseline to 12 months
Population: FGG group has 2 participants who only received FGG (n=2) and 7 participants who received FGG (n=12) and CTG at different implant sites (total of 14=2+12). CTG group has 5 participants who only received CTG (n=5) and 7 participants who received FGG and CTG (n=7) at different implant sites (total of 12=5+7).
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: implants
Arm/Group | Free Gingival Graft | Connective Tissue Graft Followed by Laser Gingivoplasty
Number analyzed (Participants) | 9 | 12
Number analyzed (implants) | 14 | 12
mm | 3.29 (1.88) | 1.29 (1.05)

2. Secondary Outcome: Measure Changes in Tissue Thickness at 2mm From GM (in mm) Between FGG and CTG
Description: Using a periodontal probe, soft tissue thickness will be measured (in mm) and compared between FGG and CTG following soft tissue grafting.
Time Frame: From baseline to 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: implant sites
Arm/Group | Free Gingival Graft | Connective Tissue Graft Followed by Laser Gingivoplasty
Number analyzed (Participants) | 9 | 12
Number analyzed (implant sites) | 14 | 12
mm | 0.21 (0.98) | 0.38 (0.8)

3. Secondary Outcome: Measure Changes in Tissue Thickness at 5mm From GM (in mm) Between FGG and CTG
Description: as for outcome 2
Time Frame: From baseline to 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: implant sites
Arm/Group | Free Gingival Graft | Connective Tissue Graft Followed by Laser Gingivoplasty
Number analyzed (Participants) | 9 | 12
Number analyzed (implant sites) | 14 | 12
mm | 0.21 (0.75) | 0.79 (0.58)

ADVERSE EVENTS:
Time Frame: from baseline through 12 months
Arm/Group | Free Gingival Graft | Connective Tissue Graft Followed by Laser Gingivoplasty | FGG + CTG
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/5 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/5 | 0/7
Other Adverse Events (participants affected / at risk) | 0/2 | 0/5 | 0/7

LIMITATIONS AND CAVEATS:
randomization was performed by site (implant) due to challenges recruiting sufficient participants for both arms

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/86/NCT03338686/Prot_SAP_000.pdf